CLINICAL TRIAL: NCT00369148
Title: Evaluation of Usefulness of Combination Therapy of Rapid Acting Insulin Secretagogue (Glinide) With Premixed Insulin in Type 2 Diabetes
Brief Title: Combination of Glinides With Premixed Insulin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Keio University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS-NHK2
Record Dates: First submitted 2006-08-28; First posted 2006-08-29 (Estimated); Last update posted 2009-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Type 2 Diabets Mellitus
Keywords: glinides; premixed insulin; combination therapy; glycemic control

INTERVENTIONS:
Drug: nateglinide(drug) mitiglinide(drug)

SUMMARY:
Combination therapy of glinides with premixed insulin provides better glycemic control than premixed insulin alone.

DETAILED DESCRIPTION:
Type 2 diabetic patients undergoing twice daily injections of premixed insulin are administered glinides (10mg of mitiglinide or 90 mg of nateglinide) at lunchtime without changing their insulin regimen. Twelve weeks after administration of the glinides, they are discontinued. HbA1c levels at the start of glinide administration, 12 weeks after administration, and 12 weeks after discontinuation are measured.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of type 2 diabetes
* Who undergoes twice daily injection of premixed insulin
* Whose HbA1c is more than 6.5% and less than 8.0%

Exclusion Criteria:

* Whose change of HbA1c is more than 1.0% during 12 weeks observational period

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2004-07; Study Completion 2006-03

PRIMARY OUTCOMES:
glycohemoglobin

SECONDARY OUTCOMES:
anhydroglucitol
lipid profile
body weight
blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Akira Shimada, MD, PhD, Study Chair — Keio University; Yoshihito Atsumi, MD, Study Director — Saiseikai Central Hospital
Locations (6):
- Japan (6):
  - Nippon Kokan Hospital, Kawasaki, Kanagawa
  - Hamamatsu Red Cross Hospital, Hamamatsu, Shizuoka
  - Saiseikai Central Hospital, Minato-ku, Tokyo
  - Kitasato Institute Hospital, Minato-ku, Tokyo
  - Keio University Hospital, Shinjuku-ku, Tokyo
  - Tokyo Metropolitan Ohtsuka Hospital, Toshima-ku, Tokyo